CLINICAL TRIAL: NCT01879878
Title: Pilot Study Evaluating Broccoli Sprouts in Advanced Pancreatic Cancer [POUDER Trial]
Acronym: POUDER
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Heidelberg University (Other)
Collaborators: German Cancer Research Center (Other)
Responsible Party: Principal Investigator, Peter Schemmer, Prof. Dr. med. Peter Schemmer, MBA, Heidelberg University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: POUDER; U1111-1144-2013 (Other: WHO)
Record Dates: First submitted 2013-06-13; First posted 2013-06-18 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2015-05

CONDITIONS: Pancreatic Ductal Adenocarcinoma
Keywords: pancreatic adenocarcinoma; broccoli sprouts; sulforaphane; palliative chemotherapy; cancer stem cells
MeSH Terms: interventions — glucoraphanin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Verum, broccoli sprout grain (Experimental): Active sulforaphane distributed in capsules each containing broccoli sprout grain
  Interventions: Dietary Supplement: Verum, broccoli sprout grain
- Placebo (Placebo Comparator): Inactive substances (methylcellulose) with identical capsule and portion distribution
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: Verum, broccoli sprout grain — Patients will be randomly classified into two groups - verum and placebo. The patients in the experimental arm will receive capsules with broccoli sprout grain containing a total of 90mg sulforaphane active substance per day over one year as nutrition supplement whereas patients assigned to the placebo group will receive inactive substance (methylcellulose) with identical capsule and portion distribution.
  Other Names: glucoraphanin
  Arms: Verum, broccoli sprout grain
Dietary Supplement: placebo — Patients assigned to the placebo group will receive inactive substance (methylcellulose) with identical capsule and portion distribution as the experimental arm.
  Arms: Placebo

SUMMARY:
The goal of the POUDER trial is to determine the feasibility of a randomized controlled trial regarding the application of freeze-dried broccoli sprouts rich in sulforaphane and quercetin in patients with advanced pancreatic ductal adenocarcinoma that receive palliative chemotherapy.

DETAILED DESCRIPTION:
Patients will be randomly classified into two groups - verum and placebo. The patients in the experimental arm will receive capsules with broccoli sprout grain containing a total of 90mg sulforaphane active substance per day over one year as nutrition supplement whereas patients assigned to the placebo group will receive inactive substance (methylcellulose) with identical capsule and portion distribution.

ELIGIBILITY:
Inclusion Criteria:

* Advanced, surgically non-treatable pancreatic ductal adenocarcinoma (surgical exploration, intraoperative biopsy but also palliative bypass interventions (bileodigestive anastomosis and/or gastroenterostomy because of preoperative cholestasis or impaired gastric emptying due to tumor-mass effect)
* Intact gastric emptying
* Written informed consent
* Patients ≥18 years of age
* Palliative chemotherapy

Exclusion Criteria:

* Intolerance to broccoli or its ingredients
* Impaired mental status or language problems / barriers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2013-12; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Feasibility of a randomized controlled trial | One year
  Main objective is to test the feasibility of a randomized controlled trial regarding the application of freeze-dried broccoli sprouts rich in sulforaphane and quercetin in patients with advanced, surgically non-resectable pancreatic ductal adenocarcinoma treated with palliative chemotherapy

SECONDARY OUTCOMES:
Disease status (imaging and tumor markers) | One year
  Disease status (cancer progress or regress): CT-imaging staging (if available) and serum tumor markers (CEA and CA-19-9) peaks as additional parameters that provide insight into disease status.

OTHER OUTCOMES:
Substance bioavailability | One year
  Urine analysis as marker of substance systemic bioavailability (conversion of the precursor glucoraphanin to the active drug substance sulforaphane). Urine analysis serves as control of the regular intake of the test substance as well.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Schemmer, Prof. Dr. med., Study Director — Heidelberg University; Ingrid Herr, Prof. Dr., Principal Investigator — Heidelberg University
Locations (1):
- Dept. of General and Transplant Surgery, University Hospital of Heidelberg, Germany, Heidelberg, Germany

REFERENCES:
- [Derived] Lozanovski VJ, Houben P, Hinz U, Hackert T, Herr I, Schemmer P. Pilot study evaluating broccoli sprouts in advanced pancreatic cancer (POUDER trial) - study protocol for a randomized controlled trial. Trials. 2014 Jun 3;15:204. doi: 10.1186/1745-6215-15-204. PMID 24894410